CLINICAL TRIAL: NCT06782256
Title: Evaluation of a Simplified Technique for Performing Laparoscopic Gastric Bypass in a Teaching Hospital
Brief Title: Simplified Technique for Performing Laparoscopic Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sandra Smith, Surgeon, Madigan Army Medical Center
Other Study IDs: 209085
Record Dates: First submitted 2010-03-08; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Gastric Bypass; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric Bypass: Patients who have undergone a laparoscopic gastric bypass procedure at using a specific surgical technique developed by the Principal Investigator

SUMMARY:
This study will include all eligible patients who have undergone or who will undergo a laparoscopic gastric bypass procedure at Madigan Army Medical Center using a specific surgical technique developed by the Principal Investigator. Traditionally, our surgeons have used a standardized technique that included use of a circular stapler to perform the anastomosis of the stomach pouch to the small bowel. The Principal Investigator developed a new technique with multiple modifications of the previous technique, including use of a totally linear stapled anastomosis. These techniques will be labeled OLD and NEW for the remainder of this document. The NEW technique was first utilized in May 2008 and has now been widely adopted by the majority of bariatric surgeons at Madigan Army Medical Center. This study will include both a retrospective review of all patients who have undergone this procedure, as well as a prospective observational study of all future patients undergoing this procedure. At this time, approximately 75 patients have undergone this procedure and will all be included in the retrospective review. The investigators estimate that 150 to 200 of these procedures will be performed at Madigan per year over the next 2 years, and will be included in the prospective observational arm of the study. The investigators anticipate a total sample number of 400 patients if the investigators collect data for the next two years.

Hypothesis: The NEW technique of gastric bypass allows for safe and rapid performance of a laparoscopic gastric bypass. The NEW technique will result in shorter operative times compared to the OLD technique, and no significant difference in postoperative complications.

DETAILED DESCRIPTION:
The methods of the retrospective arm of the study will involve abstracting of key variables of interest from review of each patient's electronic medical record, including the inpatient electronic record at the time of surgery and any subsequent readmission, and all outpatient visits identified on AHLTA. The key outcome variables of interest will be the early and late complication profile of this procedure, the impact on weight loss and control of weight-related comorbidities, the operative time required for the procedure, and the operative difficulty of the procedure as assessed by intraoperative complications and blood loss. All data will be abstracted to a standardized spreadsheet maintained by the PI, and a full listing of the study variables is attached. The prospective arm of the study will involve collection of the same data in a prospective manner, with the addition of direct conversations with the operating surgeon and/or resident to clarify any ambiguities in the electronic record.

The data analysis plan will involve simple descriptive statistics for all demographic variables, such as age, body mass index (BMI), gender, etc. Descriptive analysis of outcome data will be performed, including the short and long term complication profile of the NEW operation. Weight loss will be calculated as the percentage of the BMI lost at each time point, and will be analyzed by a paired sample t-test, with significance set at p<0.05. Operative times will be compared between different staff surgeons and different PGY levels using analysis of variance (ANOVA) with post-hoc analysis using Bonferroni test and Tamhanes T2. Complications will be compared among these same groups using chi-square analysis. As the operative times and complication profile associated with the previously performed method of gastric bypass (OLD) are known and have been published, the investigators will also compare our outcomes with this new method to our outcomes with the old method using chi-square, student's t-test, and paired t-test to compare each surgeon's operative times with the old technique and the new technique.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for a laparoscopic gastric bypass

Exclusion Criteria:

* Patients undergoing laparoscopic gastric bypass using any method other than the totally linear stapled method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone or who will undergo a laparoscopic gastric bypass procedure at Madigan Army Center using a specific surgical technique developed by the Principal Investigator.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2009-07-09 (Actual); Primary Completion 2011-03-10 (Actual); Study Completion 2011-03-10 (Actual)

PRIMARY OUTCOMES:
Complications | through study completion, an average of 2 years
  Any challenges during the procedure/operation and after

SECONDARY OUTCOMES:
Weight | through study completion, an average of 2 years
  Patient's weight
Operation Time | during surgery/procedure
  Time of operation/medical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Martin, MD, Principal Investigator — Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Background] Menifield CE, Doty N, Fletcher A. Obesity in America. ABNF J. 2008 Summer;19(3):83-8. PMID 18717205
- [Background] Drenick EJ, Bale GS, Seltzer F, Johnson DG. Excessive mortality and causes of death in morbidly obese men. JAMA. 1980 Feb 1;243(5):443-5. PMID 7351764
- [Background] Flegal KM, Graubard BI, Williamson DF, Gail MH. Cause-specific excess deaths associated with underweight, overweight, and obesity. JAMA. 2007 Nov 7;298(17):2028-37. doi: 10.1001/jama.298.17.2028. PMID 17986696
- [Background] Davis MM, Slish K, Chao C, Cabana MD. National trends in bariatric surgery, 1996-2002. Arch Surg. 2006 Jan;141(1):71-4; discussion 75. doi: 10.1001/archsurg.141.1.71. PMID 16415414
- [Background] Kinzl JF, Schrattenecker M, Traweger C, Aigner F, Fiala M, Biebl W. Quality of life in morbidly obese patients after surgical weight loss. Obes Surg. 2007 Feb;17(2):229-35. doi: 10.1007/s11695-007-9030-5. PMID 17476877
- [Background] Perry CD, Hutter MM, Smith DB, Newhouse JP, McNeil BJ. Survival and changes in comorbidities after bariatric surgery. Ann Surg. 2008 Jan;247(1):21-7. doi: 10.1097/SLA.0b013e318142cb4b. PMID 18156918
- [Background] NIH conference. Gastrointestinal surgery for severe obesity. Consensus Development Conference Panel. Ann Intern Med. 1991 Dec 15;115(12):956-61. PMID 1952493
- [Background] Shin RB. Evaluation of the learning curve for laparoscopic Roux-en-Y gastric bypass surgery. Surg Obes Relat Dis. 2005 Mar-Apr;1(2):91-4. doi: 10.1016/j.soard.2005.01.003. PMID 16925221
- [Background] Ballantyne GH, Ewing D, Capella RF, Capella JF, Davis D, Schmidt HJ, Wasielewski A, Davies RJ. The learning curve measured by operating times for laparoscopic and open gastric bypass: roles of surgeon's experience, institutional experience, body mass index and fellowship training. Obes Surg. 2005 Feb;15(2):172-82. doi: 10.1381/0960892053268507. PMID 15810124
- [Background] Gonzalez R, Lin E, Venkatesh KR, Bowers SP, Smith CD. Gastrojejunostomy during laparoscopic gastric bypass: analysis of 3 techniques. Arch Surg. 2003 Feb;138(2):181-4. doi: 10.1001/archsurg.138.2.181. PMID 12578417
- [Background] Shikora SA, Kim JJ, Tarnoff ME, Raskin E, Shore R. Laparoscopic Roux-en-Y gastric bypass: results and learning curve of a high-volume academic program. Arch Surg. 2005 Apr;140(4):362-7. doi: 10.1001/archsurg.140.4.362. PMID 15837887
- [Background] Breaux JA, Kennedy CI, Richardson WS. Advanced laparoscopic skills decrease the learning curve for laparoscopic Roux-en-Y gastric bypass. Surg Endosc. 2007 Jun;21(6):985-8. doi: 10.1007/s00464-007-9203-2. Epub 2007 Feb 16. PMID 17623252
- [Background] Hsu GP, Morton JM, Jin L, Safadi BY, Satterwhite TS, Curet MJ. Laparoscopic Roux-en-Y gastric bypass: differences in outcome between attendings and assistants of different training backgrounds. Obes Surg. 2005 Sep;15(8):1104-10. doi: 10.1381/0960892055002374. PMID 16197780
- [Background] Martin RC 2nd, Kehdy FJ, Allen JW. Formal training in advanced surgical technologies enhances the surgical residency. Am J Surg. 2005 Aug;190(2):244-8. doi: 10.1016/j.amjsurg.2005.05.020. PMID 16023439
- [Background] Madan AK, Harper JL, Tichansky DS. Techniques of laparoscopic gastric bypass: on-line survey of American Society for Bariatric Surgery practicing surgeons. Surg Obes Relat Dis. 2008 Mar-Apr;4(2):166-72; discussion 172-3. doi: 10.1016/j.soard.2007.08.006. Epub 2007 Dec 19. PMID 18069071
- [Background] Leyba JL, Llopis SN, Isaac J, Aulestia SN, Bravo C, Obregon F. Laparoscopic gastric bypass for morbid obesity-a randomized controlled trial comparing two gastrojejunal anastomosis techniques. JSLS. 2008 Oct-Dec;12(4):385-8. PMID 19275854
- [Background] Csendes A, Burgos AM, Burdiles P. Incidence of anastomotic strictures after gastric bypass: a prospective consecutive routine endoscopic study 1 month and 17 months after surgery in 441 patients with morbid obesity. Obes Surg. 2009 Mar;19(3):269-73. doi: 10.1007/s11695-008-9625-5. Epub 2008 Aug 12. PMID 18696171
- [Background] Szomstein S, Whipple OC, Zundel N, Cal P, Rosenthal R. Laparoscopic Roux-en-Y gastric bypass with linear cutter technique: comparison of four-row versus six-row cartridge in creation of anastomosis. Surg Obes Relat Dis. 2006 Jul-Aug;2(4):431-4. doi: 10.1016/j.soard.2006.03.019. PMID 16925374